CLINICAL TRIAL: NCT06621797
Title: Can L-Theanine Supplementation or Diaphragmatic Breathing Exercises in Addition to Caffeine Supplementation Be Used as Ergogenic Aids to Influence Game Performance in Esports Players?
Brief Title: Effects of Caffeine, L-Theanine, and Diaphragmatic Breathing on Esports Players' Performance
Acronym: CLD Esports St
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sedat Arslan, Assoc. Prof, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Hacettepe123; 123456789 (Other: Bandirma Onyedi Eylul University)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Esports; Caffeine; L-theanine
Keywords: Esports; Caffeine; L-Theanine; Diaphragmatic Breathing

STUDY DESIGN:
Intervention Model Description: In this randomized, single-blind crossover study, each participant will experience all three intervention conditions: (1) caffeine only, (2) caffeine combined with L-theanine, and (3) caffeine combined with diaphragmatic breathing exercises. The crossover design allows each participant to serve as their own control, reducing variability and allowing for direct comparisons between the effects of each intervention on reaction time and accuracy. Interventions are spaced apart by washout periods to ensure that the effects of one intervention do not carry over to the next. This model is ideal for studying the short-term effects of multiple interventions on esports performance.
Who Masked: Participant
Masking Description: In this study, participants are masked to the specific intervention they are receiving during each phase. They are unaware of whether they are receiving caffeine only, caffeine combined with L-theanine, or caffeine combined with diaphragmatic breathing exercises. The researcher administering the interventions and conducting assessments is aware of the interventions, ensuring that the study remains single-blind. No other parties are masked in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeine Only Arm (Experimental): Participants receive a caffeine supplement only.
  Interventions: Dietary Supplement: Intervention 1: Dietary Supplement - Caffeine Supplement
- Caffeine + L-Theanine Arm (Experimental): Participants receive a combination of caffeine and L-theanine supplements.
  Interventions: Dietary Supplement: Intervention 2: Dietary Supplement - Caffeine + L-Theanine Supplement
- Caffeine + Diaphragmatic Breathing Exercises Arm (Experimental): Participants receive a caffeine supplement and perform diaphragmatic breathing exercises.
  Interventions: Behavioral: Intervention 3: Dietary Supplement - Caffeine Supplement + Diaphragmatic Breathing Exercises

INTERVENTIONS:
Dietary Supplement: Intervention 1: Dietary Supplement - Caffeine Supplement — Participants in this group will receive a caffeine supplement (3 mg/kg body weight) taken orally 45 minutes before performance testing. No additional interventions will be administered.
  Arms: Caffeine Only Arm
Dietary Supplement: Intervention 2: Dietary Supplement - Caffeine + L-Theanine Supplement — Participants in this group will receive a caffeine supplement (3 mg/kg body weight) along with L-theanine in a 1:2 ratio taken orally 45 minutes before performance testing.
  Arms: Caffeine + L-Theanine Arm
Behavioral: Intervention 3: Dietary Supplement - Caffeine Supplement + Diaphragmatic Breathing Exercises — Participants in this group will receive a caffeine supplement (3 mg/kg body weight) 45 minutes before performance testing, followed by a 10-minute session of diaphragmatic breathing exercises.
  Arms: Caffeine + Diaphragmatic Breathing Exercises Arm

SUMMARY:
The purpose of this study is to investigate whether caffeine, L-theanine (a natural amino acid found in tea), and diaphragmatic breathing exercises can help improve the game performance of esports players. Esports players often need fast reaction times, high accuracy, and mental focus during competitive gaming. This study will look at how caffeine and L-theanine supplements, either separately or together, and breathing exercises impact key performance factors like reaction time and accuracy during gameplay. The goal is to determine if these strategies can help esports players perform better by reducing stress, improving concentration, and speeding up reaction times. The findings could help inform safe, effective methods to enhance cognitive and physical performance in gaming.

DETAILED DESCRIPTION:
This study explores the effects of caffeine, L-theanine supplementation, and diaphragmatic breathing exercises on esports players' game performance, focusing on reaction time and accuracy. Caffeine is widely recognized for its stimulating effects, improving attention and reducing fatigue, while L-theanine, found in tea, is known to reduce stress and balance the effects of caffeine. Diaphragmatic breathing exercises are designed to lower stress levels, improve focus, and enhance cognitive function.

The study utilizes a randomized, single-blind crossover design, where participants-esports players aged 18-30-will undergo three different interventions: caffeine only, caffeine combined with L-theanine, and caffeine combined with diaphragmatic breathing exercises. Performance outcomes, including reaction time and accuracy, will be assessed using game-based software and tests. Participants will have their performance measured before and after each intervention, allowing for comparison between the different strategies.

This study aims to determine whether these supplements and exercises, alone or in combination, can serve as effective ergogenic aids, helping esports players optimize their performance by improving cognitive and motor skills, while also reducing stress. These findings could have broader applications for enhancing mental performance in competitive environments.

ELIGIBILITY:
Inclusion Criteria:

* Male esports players aged 18-30.
* Actively involved in esports for at least 6 hours per week for a minimum of 6 months.
* Low caffeine consumption (less than 80 mg per day).
* Low L-theanine consumption (less than 100 mg per day).
* Non-smokers or those who do not use tobacco products.
* No recent history of upper extremity surgery.
* No known allergies to caffeine or L-theanine.
* No neurological, visual, or auditory disorders.
* No use of drugs or performance-enhancing supplements within the past month.
* No alcohol consumption within the past week.

Exclusion Criteria:

* Use of stimulant medications.
* History of upper extremity surgery.
* Diagnosed neurological, visual, or auditory disorders.
* Allergy to caffeine or L-theanine.
* Use of drugs or performance-enhancing supplements within the past month.
* Regular tobacco use.
* Consumption of alcohol in the past week.
* Inconsistent sleep patterns or difficulty following standardized sleep and hydration guidelines.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male participants only are eligible to participate in this study, as all participants will be male esports players aged 18-30, based on the inclusion criteria specified.
Enrollment: 15 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Reaction Time | Reaction time will be assessed immediately before each intervention and at two time points after each intervention (at 45 minutes and 2 hours post-intervention) on each of the three study days.
  The time it takes for participants to respond to visual and auditory stimuli during gaming, measured in milliseconds using Aim Lab and other standardized reaction time tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, there is no plan to share IPD with other researchers.